CLINICAL TRIAL: NCT03078166
Title: Global Congestive Heart Failure Registry
Acronym: G-CHF
Status: Completed | Type: Observational
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Population Health Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 0812
Record Dates: First submitted 2017-03-07; First posted 2017-03-13 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Heart Failure
Keywords: Cardiac Failure; Congestive Heart Failure; Heart Decompensation; Heart Failure, Congestive; Heart Failure, Left-Sided; Heart Failure, Right-Sided; Left-Sided Heart Failure; Myocardial Failure; Right-Sided Heart Failure; Outcomes; Co-morbidities; Biomarkers
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Approximately 4000 patients (a subset of the main G-CHF study population) will have blood and urine collected. Anonymized specimens will be sent to a central laboratory in Hamilton, Ontario, Canada for further storage and analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Heart failure (HF) is a major health problem worldwide but there is no global HF study that documents demographics, socioeconomic and clinical factors, diagnostic and management patterns, etiology, biomarkers, co-morbidities, treatments, quality of life, barriers to care and outcomes in all parts of the world. Such knowledge is essential in the prevention and treatment of this global disease. The Global Congestive Heart Failure Registry (G-CHF) is a global registry of approximately 20,000-25,000 HF patients enrolled over approximately 5 years to study these risks and causes of HF.

DETAILED DESCRIPTION:
The G-CHF Registry is a prospective global cohort study of approximately 20,000-25,000 HF patients enrolled over approximately 5 years. Baseline data will be obtained on demographic and socioeconomic data, clinical and laboratory variables, co-morbidities, biomarkers, echocardiography, HF causes, medication use, management patterns, quality of life, and health systems. Six-month, 12-month, 18-month and 24-month follow-up data will be obtained to document patient outcomes and factors associated with outcomes.

A sub-study of approximately 4000 patients (a subset of the main study population) will be performed to measure frailty, cognitive and lung function, mental health, medication adherence, patient-reported barriers to care, dietary assessment, and collection of blood and urine samples for central storage and analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age with a clinical diagnosis of HF seen in outpatient clinics or inpatient hospital wards of the participating centres.
* Written informed consent

Exclusion Criteria:

* Patients considered unreliable by the investigator concerning the requirements for follow-up visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HF will be recruited from approximately 200-300 centers in North America, South America, Europe, Africa, Asia, the Middle East, and Australia over approximately 5 years (approximately 4,000-5,000 patients per year), resulting in an initial sample estimate of approximately 20,000-25,000 patients. In each country, approximately 2/3 of patients will be recruited from the outpatient clinic setting (chronic HF) and 1/3 from the hospital inpatient setting (acute HF or acute exacerbation of chronic HF). At least one site in each country will be rural.
Sampling Method: Non-Probability Sample
Enrollment: 25000 (Estimated)
Dates: Start 2016-12-20 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Mortality, by cause | 2 years
  The main objective of G-CHF is to obtain reliable estimates of mortality and other non-fatal clinical outcomes in HF patients overall and in 6 global regions. Factors associated with outcomes will be explored. All outcome events will be recorded and summarized individually as rates and proportions, with two-sided confidence intervals calculated.

SECONDARY OUTCOMES:
Non-fatal major clinical events (both resulting in and not resulting in hospitalization) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Salim Yusuf, DPhil, FRCPC, FRSC, O.C., Principal Investigator — Executive Director; Hisham Dokainish, M.D., FRCPC, FASE, FACC, Principal Investigator — Internal PHRI Lead Investigator
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Johansson I, Joseph P, Balasubramanian K, McMurray JJV, Lund LH, Ezekowitz JA, Kamath D, Alhabib K, Bayes-Genis A, Budaj A, Dans ALL, Dzudie A, Probstfield JL, Fox KAA, Karaye KM, Makubi A, Fukakusa B, Teo K, Temizhan A, Wittlinger T, Maggioni AP, Lanas F, Lopez-Jaramillo P, Silva-Cardoso J, Sliwa K, Dokainish H, Grinvalds A, McCready T, Yusuf S; G-CHF Investigators. Health-Related Quality of Life and Mortality in Heart Failure: The Global Congestive Heart Failure Study of 23 000 Patients From 40 Countries. Circulation. 2021 Jun;143(22):2129-2142. doi: 10.1161/CIRCULATIONAHA.120.050850. Epub 2021 Apr 28. PMID 33906372